CLINICAL TRIAL: NCT04210557
Title: Models of Auditory Hallucination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough suitable participants.
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2000023640; 1R21MH116258-01A1 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-12-24 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia; Schizo Affective Disorder; Auditory Hallucination
Keywords: TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participant, the physician administering TMS, and the research psychologist will be blind to the condition. One research assistant will be unblinded to the condition. This unblinded research assistant is responsible for setting up the active TMS coils or the sham TMS coils and determining the protocol used, to maintain the blindness of other study staff and the participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS to insula (Active Comparator): This study will recruit 30 clinical voice hearers (P+H+). They will complete two parallel forms of the conditioned hallucinations task (with different visual and auditory stimuli) on two occasions, separated by a week.
  TMS and sham will be delivered in a randomized counterbalanced order. Hypothesis: Inhibiting the insula will decrease prior over-weighting. If this computational perturbation is responsible for conditioned hallucinations, then ameliorating it with TMS that increases insula engagement will decrease conditioned hallucination responses. Furthermore, the prior weighting parameter will be reduced following active TMS compared with sham.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS to cerebellum (Active Comparator): This study will recruit a further 70 clinical voice hearers. Again, they will complete parallel forms of the conditioned hallucinations task on two occasions, separated by a week. They will receive excitatory TMS over the cerebellum (and sham on the other occasion, in a randomized counterbalanced order). Hypotheses: Exciting the cerebellum will increase belief-updating. If poor belief-updating contributes to conditioned hallucinations, increasing cerebellum engagement should decrease conditioned hallucinations and alter the belief-updating model parameter compared with sham TMS.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction. An electric pulse generator, or stimulator, is connected to a magnetic coil, which in turn is connected to the scalp. The stimulator generates a changing electric current within the coil which induces a magnetic field; this field then causes a second inductance of inverted electric charge within the brain itself.
  Other Names: repetitive transcranial magnetic stimulation (rTMS)

SUMMARY:
The purpose of this study is to address the shortcoming in clinical hallucination research by causally manipulating the neural loci of conditioned hallucination task behavior in-person in patients with psychosis using transcranial magnetic stimulation (TMS), tracking the impact of this manipulation on the number of times participants with hallucinations report hearing tones that were not presented. With such a causal intervention, the veracity of this explanation of hallucinations will be either validated or disconfirmed. If validated, the task can be further developed as a biomarker for predicting the hallucination onset, guiding, developing or tracking the effects of treatments for hallucinations.

DETAILED DESCRIPTION:
Hallucinations are percepts without stimulus. 70% of patients with schizophrenia suffer distressing auditory hallucinations. Their mere presence increases the risk of suicide. Most reach remission with D2 dopamine receptor blocking drugs after 1 year of adherence. However, 30% of patients have intractable hallucinations, and 50% are non-adherent to their medications, commonly because of unfavorable side-effects - those intractable and non-adherent patients continue to suffer. There is a clear need for a mechanistic understanding of hallucinations as a prelude to rational treatment design.

This study provides the initial steps towards the development of an interventional biomarker for clinical hallucinations, grounded in computational neuroscience.

Computational psychiatry involves harnessing the power of computational neuroscience to address the clinical needs of those suffering from serious mental illnesses. There has been much discussion of the promise of the approach. There have been few studies thus far and they have largely involved correlative methods like functional neuroimaging. This study will address this shortcoming by causally manipulating the neural loci of computational model parameters in-person in patients with psychosis using transcranial magnetic stimulation (TMS), tracking the impact of this manipulation on behavioral task performance . With such a causal intervention, the veracity of the model's explanation of hallucinations will be either validated or disconfirmed. If validated, the model can be further developed as a biomarker for predicting the hallucination onset, guiding, developing or tracking the effects of treatments for hallucinations. If disconfirmed, the model ought to be discarded and other alternatives should be pursued.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 45 years
* Voice hearing patients
* Meet diagnostic criteria for DSM-V schizophrenia or schizophreniform disorder
* Report hearing voices at least once a day
* Score > 3 on PANSS P3 (hallucinations item)

Exclusion Criteria:

* DSM-V substance use disorder within the past 6 months
* Previous head injury with neurological symptoms and/or unconsciousness
* Intellectual disability (IQ < 70)
* Non-English speaker
* Contraindications for TMS, including:

  * History of seizures
  * Metallic implants
  * Pacemaker
  * Pregnancy
* Less than 6 weeks of a stable dose of psychotropic medication(s)
* Comorbid mood or anxiety diagnosis
* Clinically/behaviorally instability and unable to cooperate with TMS procedures
* Clinically significant medical condition(s)
* Unstable medical condition(s) based on EKG, medical history, physical examination, and routine lab work
* Personal history of stroke
* Family history of seizures

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Corlett, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center (CMHC), New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pompili M, Amador XF, Girardi P, Harkavy-Friedman J, Harrow M, Kaplan K, Krausz M, Lester D, Meltzer HY, Modestin J, Montross LP, Mortensen PB, Munk-Jorgensen P, Nielsen J, Nordentoft M, Saarinen PI, Zisook S, Wilson ST, Tatarelli R. Suicide risk in schizophrenia: learning from the past to change the future. Ann Gen Psychiatry. 2007 Mar 16;6:10. doi: 10.1186/1744-859X-6-10. PMID 17367524
- [Background] Kelleher I, Lynch F, Harley M, Molloy C, Roddy S, Fitzpatrick C, Cannon M. Psychotic symptoms in adolescence index risk for suicidal behavior: findings from 2 population-based case-control clinical interview studies. Arch Gen Psychiatry. 2012 Dec;69(12):1277-83. doi: 10.1001/archgenpsychiatry.2012.164. PMID 23108974
- [Background] Harkavy-Friedman JM, Kimhy D, Nelson EA, Venarde DF, Malaspina D, Mann JJ. Suicide attempts in schizophrenia: the role of command auditory hallucinations for suicide. J Clin Psychiatry. 2003 Aug;64(8):871-4. PMID 12927000
- [Background] Friston K. Hierarchical models in the brain. PLoS Comput Biol. 2008 Nov;4(11):e1000211. doi: 10.1371/journal.pcbi.1000211. Epub 2008 Nov 7. PMID 18989391
- [Background] Friston K. The free-energy principle: a rough guide to the brain? Trends Cogn Sci. 2009 Jul;13(7):293-301. doi: 10.1016/j.tics.2009.04.005. Epub 2009 Jun 24. PMID 19559644
- [Background] Powers AR, Mathys C, Corlett PR. Pavlovian conditioning-induced hallucinations result from overweighting of perceptual priors. Science. 2017 Aug 11;357(6351):596-600. doi: 10.1126/science.aan3458. PMID 28798131
- [Background] Powers AR III, Kelley M, Corlett PR. Hallucinations as top-down effects on perception. Biol Psychiatry Cogn Neurosci Neuroimaging. 2016 Sep;1(5):393-400. doi: 10.1016/j.bpsc.2016.04.003. PMID 28626813
- [Background] Helmholtz, H., & Southall, J. P. C. (1924). Helmholtz's treatise on physiological optics. Rochester, N.Y.: Optical Society of America.
- [Background] Friston K. A theory of cortical responses. Philos Trans R Soc Lond B Biol Sci. 2005 Apr 29;360(1456):815-36. doi: 10.1098/rstb.2005.1622. PMID 15937014
- [Background] Rao RP, Ballard DH. Predictive coding in the visual cortex: a functional interpretation of some extra-classical receptive-field effects. Nat Neurosci. 1999 Jan;2(1):79-87. doi: 10.1038/4580. PMID 10195184
- [Background] Bayes T. An essay towards solving a problem in the doctrine of chances. 1763. MD Comput. 1991 May-Jun;8(3):157-71. No abstract available. PMID 1857193
- [Background] Adams RA, Stephan KE, Brown HR, Frith CD, Friston KJ. The computational anatomy of psychosis. Front Psychiatry. 2013 May 30;4:47. doi: 10.3389/fpsyt.2013.00047. eCollection 2013. PMID 23750138
- [Background] Friston, K. (2005). Hallucinations and perceptual inference. Behavioral and Brain Sciences, 28(6), 764-766. doi:10.1017/S0140525X05290131
- [Background] G. Ellson, D. (1941). Hallucinations produced by sensory conditioning. Journal of Experimental Psychology. 28. 1-20. 10.1037/h0054167.
- [Background] Mathys C, Daunizeau J, Friston KJ, Stephan KE. A bayesian foundation for individual learning under uncertainty. Front Hum Neurosci. 2011 May 2;5:39. doi: 10.3389/fnhum.2011.00039. eCollection 2011. PMID 21629826
- [Background] Watson AB, Pelli DG. QUEST: a Bayesian adaptive psychometric method. Percept Psychophys. 1983 Feb;33(2):113-20. doi: 10.3758/bf03202828. No abstract available. PMID 6844102
- [Background] Verdoux H, van Os J. Psychotic symptoms in non-clinical populations and the continuum of psychosis. Schizophr Res. 2002 Mar 1;54(1-2):59-65. doi: 10.1016/s0920-9964(01)00352-8. PMID 11853979
- [Background] Powers AR 3rd, Kelley MS, Corlett PR. Varieties of Voice-Hearing: Psychics and the Psychosis Continuum. Schizophr Bull. 2017 Jan;43(1):84-98. doi: 10.1093/schbul/sbw133. Epub 2016 Oct 7. PMID 28053132
- [Background] Zmigrod L, Garrison JR, Carr J, Simons JS. The neural mechanisms of hallucinations: A quantitative meta-analysis of neuroimaging studies. Neurosci Biobehav Rev. 2016 Oct;69:113-23. doi: 10.1016/j.neubiorev.2016.05.037. Epub 2016 Jul 26. PMID 27473935
- [Background] Mathys CD, Lomakina EI, Daunizeau J, Iglesias S, Brodersen KH, Friston KJ, Stephan KE. Uncertainty in perception and the Hierarchical Gaussian Filter. Front Hum Neurosci. 2014 Nov 19;8:825. doi: 10.3389/fnhum.2014.00825. eCollection 2014. PMID 25477800
- [Background] Guediche S, Holt LL, Laurent P, Lim SJ, Fiez JA. Evidence for Cerebellar Contributions to Adaptive Plasticity in Speech Perception. Cereb Cortex. 2015 Jul;25(7):1867-77. doi: 10.1093/cercor/bht428. Epub 2014 Jan 22. PMID 24451660
- [Background] Shergill SS, White TP, Joyce DW, Bays PM, Wolpert DM, Frith CD. Functional magnetic resonance imaging of impaired sensory prediction in schizophrenia. JAMA Psychiatry. 2014 Jan;71(1):28-35. doi: 10.1001/jamapsychiatry.2013.2974. PMID 24196370
- [Background] George MS. Stimulating the brain. Sci Am. 2003 Sep;289(3):66-73. doi: 10.1038/scientificamerican0903-66. No abstract available. PMID 12951829
- [Background] Hoffman RE, Boutros NN, Berman RM, Roessler E, Belger A, Krystal JH, Charney DS. Transcranial magnetic stimulation of left temporoparietal cortex in three patients reporting hallucinated "voices". Biol Psychiatry. 1999 Jul 1;46(1):130-2. doi: 10.1016/s0006-3223(98)00358-8. PMID 10394483
- [Background] Kring AM, Gur RE, Blanchard JJ, Horan WP, Reise SP. The Clinical Assessment Interview for Negative Symptoms (CAINS): final development and validation. Am J Psychiatry. 2013 Feb;170(2):165-72. doi: 10.1176/appi.ajp.2012.12010109. PMID 23377637
- [Background] Borckardt JJ, Nahas Z, Koola J, George MS. Estimating resting motor thresholds in transcranial magnetic stimulation research and practice: a computer simulation evaluation of best methods. J ECT. 2006 Sep;22(3):169-75. doi: 10.1097/01.yct.0000235923.52741.72. PMID 16957531
- [Background] Arana AB, Borckardt JJ, Ricci R, Anderson B, Li X, Linder KJ, Long J, Sackeim HA, George MS. Focal electrical stimulation as a sham control for repetitive transcranial magnetic stimulation: Does it truly mimic the cutaneous sensation and pain of active prefrontal repetitive transcranial magnetic stimulation? Brain Stimul. 2008 Jan;1(1):44-51. doi: 10.1016/j.brs.2007.08.006. PMID 19424459
- [Background] Stromer R, McIlvane W.J, Serna R.W. Complex stimulus control and equivalence. The Psychological Record. 1993;43:585-598.
- [Background] Gekas N, Chalk M, Seitz AR, Series P. Complexity and specificity of experimentally-induced expectations in motion perception. J Vis. 2013 Mar 13;13(4):8. doi: 10.1167/13.4.8. PMID 23487160
- [Background] Jones PD, Holding DH. Extremely long-term persistence of the McCollough effect. J Exp Psychol Hum Percept Perform. 1975 Nov;1(4):323-7. doi: 10.1037//0096-1523.1.4.323. PMID 1185119
- [Background] Shams L, Seitz AR. Benefits of multisensory learning. Trends Cogn Sci. 2008 Nov;12(11):411-7. doi: 10.1016/j.tics.2008.07.006. PMID 18805039
- [Background] Downar J, Blumberger DM, Daskalakis ZJ. The Neural Crossroads of Psychiatric Illness: An Emerging Target for Brain Stimulation. Trends Cogn Sci. 2016 Feb;20(2):107-120. doi: 10.1016/j.tics.2015.10.007. Epub 2015 Dec 3. PMID 26655436
- [Background] Dinur-Klein L, Dannon P, Hadar A, Rosenberg O, Roth Y, Kotler M, Zangen A. Smoking cessation induced by deep repetitive transcranial magnetic stimulation of the prefrontal and insular cortices: a prospective, randomized controlled trial. Biol Psychiatry. 2014 Nov 1;76(9):742-9. doi: 10.1016/j.biopsych.2014.05.020. Epub 2014 Jun 5. PMID 25038985
- [Background] Hardwick RM, Lesage E, Miall RC. Cerebellar transcranial magnetic stimulation: the role of coil geometry and tissue depth. Brain Stimul. 2014 Sep-Oct;7(5):643-9. doi: 10.1016/j.brs.2014.04.009. Epub 2014 May 6. PMID 24924734
- [Background] Demirtas-Tatlidede A, Freitas C, Cromer JR, Safar L, Ongur D, Stone WS, Seidman LJ, Schmahmann JD, Pascual-Leone A. Safety and proof of principle study of cerebellar vermal theta burst stimulation in refractory schizophrenia. Schizophr Res. 2010 Dec;124(1-3):91-100. doi: 10.1016/j.schres.2010.08.015. PMID 20817483
- [Background] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Background] Rosner, B. Fundamentals of biostatistics. 1995. Duxbury Press: New York.
- [Background] Gulli G, Tarperi C, Cevese A, Acler M, Bongiovanni G, Manganotti P. Effects of prefrontal repetitive transcranial magnetic stimulation on the autonomic regulation of cardiovascular function. Exp Brain Res. 2013 Apr;226(2):265-71. doi: 10.1007/s00221-013-3431-6. Epub 2013 Mar 2. PMID 23455721
- [Background] Kimhy D, Wall MM, Hansen MC, Vakhrusheva J, Choi CJ, Delespaul P, Tarrier N, Sloan RP, Malaspina D. Autonomic Regulation and Auditory Hallucinations in Individuals With Schizophrenia: An Experience Sampling Study. Schizophr Bull. 2017 Jul 1;43(4):754-763. doi: 10.1093/schbul/sbw219. PMID 28177507
- [Background] Flashman LA, Flaum M, Gupta S, Andreasen NC. Soft signs and neuropsychological performance in schizophrenia. Am J Psychiatry. 1996 Apr;153(4):526-32. doi: 10.1176/ajp.153.4.526. PMID 8599401
- [Background] Miall RC, Christensen LO. The effect of rTMS over the cerebellum in normal human volunteers on peg-board movement performance. Neurosci Lett. 2004 Nov 23;371(2-3):185-9. doi: 10.1016/j.neulet.2004.08.067. PMID 15519754
- [Background] Davies P, Davies GL, Bennett S. An effective paradigm for conditioning visual perception in human subjects. Perception. 1982;11(6):663-9. doi: 10.1068/p110663. PMID 7186617
- [Background] Dobek CE, Blumberger DM, Downar J, Daskalakis ZJ, Vila-Rodriguez F. Risk of seizures in transcranial magnetic stimulation: a clinical review to inform consent process focused on bupropion. Neuropsychiatr Dis Treat. 2015 Nov 30;11:2975-87. doi: 10.2147/NDT.S91126. eCollection 2015. PMID 26664122
- [Background] Maizey L, Allen CP, Dervinis M, Verbruggen F, Varnava A, Kozlov M, Adams RC, Stokes M, Klemen J, Bungert A, Hounsell CA, Chambers CD. Comparative incidence rates of mild adverse effects to transcranial magnetic stimulation. Clin Neurophysiol. 2013 Mar;124(3):536-44. doi: 10.1016/j.clinph.2012.07.024. Epub 2012 Sep 15. PMID 22986284
- [Background] Anderson BS, Kavanagh K, Borckardt JJ, Nahas ZH, Kose S, Lisanby SH, McDonald WM, Avery D, Sackeim HA, George MS. Decreasing procedural pain over time of left prefrontal rTMS for depression: initial results from the open-label phase of a multi-site trial (OPT-TMS). Brain Stimul. 2009 Apr;2(2):88-92. doi: 10.1016/j.brs.2008.09.001. PMID 20161310
- [Background] Pascual-Leone A, Houser CM, Reese K, Shotland LI, Grafman J, Sato S, Valls-Sole J, Brasil-Neto JP, Wassermann EM, Cohen LG, et al. Safety of rapid-rate transcranial magnetic stimulation in normal volunteers. Electroencephalogr Clin Neurophysiol. 1993 Apr;89(2):120-30. doi: 10.1016/0168-5597(93)90094-6. PMID 7683602
- [Background] Horwitz NH. Historical perspective. David Ferrier (1843-1928). Neurosurgery. 1994 Oct;35(4):793-5. doi: 10.1227/00006123-199410000-00042. No abstract available. PMID 7808632
- [Background] Morabito C. David Ferrier and Luigi Luciani on the localization of brain functions. Physis Riv Int Stor Sci. 1999;36(2):387-405. PMID 11640241
- [Background] Bohning, D. E. (2000). Introduction and overview of TMS physics. Transcranial magnetic stimulation in neuropsychiatry, 13-44.
- [Background] George MS, Aston-Jones G. Noninvasive techniques for probing neurocircuitry and treating illness: vagus nerve stimulation (VNS), transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS). Neuropsychopharmacology. 2010 Jan;35(1):301-16. doi: 10.1038/npp.2009.87. PMID 19693003
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] Johnson KA, Baig M, Ramsey D, Lisanby SH, Avery D, McDonald WM, Li X, Bernhardt ER, Haynor DR, Holtzheimer PE 3rd, Sackeim HA, George MS, Nahas Z. Prefrontal rTMS for treating depression: location and intensity results from the OPT-TMS multi-site clinical trial. Brain Stimul. 2013 Mar;6(2):108-17. doi: 10.1016/j.brs.2012.02.003. Epub 2012 Mar 14. PMID 22465743
- [Background] Janicak PG, Nahas Z, Lisanby SH, Solvason HB, Sampson SM, McDonald WM, Marangell LB, Rosenquist P, McCall WV, Kimball J, O'Reardon JP, Loo C, Husain MH, Krystal A, Gilmer W, Dowd SM, Demitrack MA, Schatzberg AF. Durability of clinical benefit with transcranial magnetic stimulation (TMS) in the treatment of pharmacoresistant major depression: assessment of relapse during a 6-month, multisite, open-label study. Brain Stimul. 2010 Oct;3(4):187-99. doi: 10.1016/j.brs.2010.07.003. Epub 2010 Aug 11. PMID 20965447
- [Background] Mantovani A, Pavlicova M, Avery D, Nahas Z, McDonald WM, Wajdik CD, Holtzheimer PE 3rd, George MS, Sackeim HA, Lisanby SH. Long-term efficacy of repeated daily prefrontal transcranial magnetic stimulation (TMS) in treatment-resistant depression. Depress Anxiety. 2012 Oct;29(10):883-90. doi: 10.1002/da.21967. Epub 2012 Jun 11. PMID 22689290
- [Background] Carpenter LL, Janicak PG, Aaronson ST, Boyadjis T, Brock DG, Cook IA, Dunner DL, Lanocha K, Solvason HB, Demitrack MA. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of acute treatment outcomes in clinical practice. Depress Anxiety. 2012 Jul;29(7):587-96. doi: 10.1002/da.21969. Epub 2012 Jun 11. PMID 22689344
- [Background] Hoffman RE, Wu K, Pittman B, Cahill JD, Hawkins KA, Fernandez T, Hannestad J. Transcranial magnetic stimulation of Wernicke's and Right homologous sites to curtail "voices": a randomized trial. Biol Psychiatry. 2013 May 15;73(10):1008-14. doi: 10.1016/j.biopsych.2013.01.016. Epub 2013 Feb 26. PMID 23485015
- [Background] Chen R, Gerloff C, Classen J, Wassermann EM, Hallett M, Cohen LG. Safety of different inter-train intervals for repetitive transcranial magnetic stimulation and recommendations for safe ranges of stimulation parameters. Electroencephalogr Clin Neurophysiol. 1997 Dec;105(6):415-21. doi: 10.1016/s0924-980x(97)00036-2. PMID 9448642
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Anderson B, Mishory A, Nahas Z, Borckardt JJ, Yamanaka K, Rastogi K, George MS. Tolerability and safety of high daily doses of repetitive transcranial magnetic stimulation in healthy young men. J ECT. 2006 Mar;22(1):49-53. doi: 10.1097/00124509-200603000-00011. PMID 16633208
- [Background] Rachid F. Maintenance repetitive transcranial magnetic stimulation (rTMS) for relapse prevention in with depression: A review. Psychiatry Res. 2018 Apr;262:363-372. doi: 10.1016/j.psychres.2017.09.009. Epub 2017 Sep 19. PMID 28951141

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS to Insula: This study will recruit 30 clinical voice hearers (P+H+). They will complete two parallel forms of the conditioned hallucinations task (with different visual and auditory stimuli) on two occasions, separated by a week.
  TMS and sham will be delivered in a randomized counterbalanced order. Hypothesis: Inhibiting the insula will decrease prior over-weighting. If this computational perturbation is responsible for conditioned hallucinations, then ameliorating it with TMS that increases insula engagement will decrease conditioned hallucination responses. Furthermore, the prior weighting parameter will be reduced following active TMS compared with sham.
  Transcranial Magnetic Stimulation (TMS): Transcranial magnetic stimulation (TMS) is a noninvasive form of brain stimulation in which a changing magnetic field is used to cause electric current at a specific area of the brain through electromagnetic induction. An electric pulse generator, or stimulator, is connected to a magnetic coil, which in turn is connected to the scalp. The stimulator generates a changing electric current within the coil which induces a magnetic field; this field then causes a second inductance of inverted electric charge within the brain itself.
Period: Overall Study
Arm/Group | TMS to Insula | TMS to Cerebellum
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data not reported to avoid making any identifying characteristics public.
Groups:
- Total: Total of all reporting groups
Arm/Group | TMS to Insula | TMS to Cerebellum | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Conditioned Hallucinations Task Performance
Description: The primary outcome measure is the number of times participants report hearing tones that were not presented. There are 360 total trials. There are 120 no tone trials. People who hear voices typically report hearing tones on 30% of the no tone trials (approximately 36 times, as compared to 12 times in people who do not hear voices). The investigators anticipate fewer conditioned hallucinations (fewer than 36 reports of tones when none were presented) in the active TMS conditions as compared to the sham.
Time Frame: approximately 13 months
Population: Data not reported to avoid making any identifying characteristics public.
Arm/Group | TMS to Insula | TMS to Cerebellum
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: approximately 13 months
Description: Zero at risk because 0 were enrolled in that arm.
Arm/Group | TMS to Insula | TMS to Cerebellum
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04210557/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT04210557/ICF_001.pdf